CLINICAL TRIAL: NCT01515384
Title: A Preliminary Evaluation of the Safety and Pancreas Imaging Properties of 18F-AV-133 in Healthy Volunteers and in Patients With Type 1 or Type 2 Diabetes
Brief Title: A Trial of 18F-AV-133 Positron Emission Tomography (PET)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-133-D01
Record Dates: First submitted 2011-02-21; First posted 2012-01-24 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — florbenazine F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Type 1 Diabetes (Experimental)
  Interventions: Drug: 18F-AV-133
- Type 2 Diabetes (Experimental)
  Interventions: Drug: 18F-AV-133
- Healthy Controls (Experimental)
  Interventions: Drug: 18F-AV-133

INTERVENTIONS:
Drug: 18F-AV-133 — IV injection, 7.6 mCi (281.2 MBq)

SUMMARY:
The purpose of this study is to evaluate the safety and pancreas imaging properties of 18F-AV-133.

DETAILED DESCRIPTION:
The primary objective of this protocol is to address the feasibility for further development of the VMAT2-binding compound 18F-AV-133 as a diagnostic radiopharmaceutical in the field of diabetes. Specifically, this study will evaluate 18F-AV-133 imaging in patients with type 1 diabetes, patients with type 2 diabetes and in healthy controls in order to:

1. Obtain information regarding the safety of 18F-AV-133 in these populations;
2. Determine whether uptake, distribution, or clearance of 18F-AV-133 in the pancreas differs between subjects with predicted reduced beta cell mass (patients with type 1 or type 2 diabetes of long duration) and normal beta cell mass (healthy volunteers);
3. Evaluate the PET imaging pharmacokinetics of 18F-AV-133 in abdominal organs of healthy control subjects and patients with type 1 or type 2 diabetes;
4. Obtain preliminary information regarding the appropriate time window for optimal PET imaging of 18F-AV-133 in the pancreas post-administration for type 1, type 2, and normal healthy individuals;
5. Obtain preliminary information regarding an appropriate reference tissue for evaluating the PET imaging results of 18F-AV-133 in the pancreas; and
6. Evaluate the imaging properties of 18F-AV-133 in the pancreas relative to the brain in a subset of subjects.

ELIGIBILITY:
Patients with type 1 diabetes may be enrolled if they meet all of the following criteria:

* Are males or females between 18 and 70 years of age, inclusive;
* Have a diagnosis of type 1 diabetes mellitus as defined by ADA criteria; diabetes onset younger than age 21, duration >5 years; Insulin dose requirements ≤ 0.8 units/kg/day;
* HbA1c level ≥ 5% and ≤ 8%;
* Have fasting C-Peptide < 0.1 ng/ml;
* Have a BMI between 18 and 32 kg/m2;
* Able to tolerate PET imaging;
* In the judgment of the physician, are capable of fasting 4-6 hours prior to screening and Day 1 imaging procedures; and
* Give informed consent.

Patients with type 2 diabetes may be enrolled if they meet all of the following criteria:

* Are males or females between 18 and 70 years of age, inclusive;
* Must have been diagnosed with type 2 diabetes for more than five years;
* HbA1c level ≥ 5% and ≤ 8%;
* Have a BMI between 18 and 32 kg/m2;
* Glucose > 200 mg/dl on Mixed Meal Tolerance Test at screening visit;
* Able to tolerate PET imaging;
* In the judgment of the physician, are capable of fasting 4-6 hours prior to screening and Day 1 imaging procedures; and
* Give informed consent.

Healthy volunteers may be enrolled if they meet all of the following criteria:

* Are males or females between 18 and 70 years of age, inclusive;
* Have no history of type 1 or type 2 diabetes in a first degree relative;
* Fasting blood glucose ≤ 100 mg/dL;
* HbA1c level ≤ 6%;
* Normal Mixed Meal Tolerance test at screening visit;
* BMI between 18 and 32 kg/m2;
* Able to tolerate PET imaging;
* In the judgment of the physician, are capable of fasting 4-6 hours prior to screening and Day 1 imaging procedures; and
* Give informed consent.

Subjects will be excluded from enrollment if they meet any of the following criteria:

* Clinically significant renal dysfunction;
* Clinically significant liver dysfunction as determined by history, physical examination, and standard liver function testing at screening (AST, ALT, Total/Direct Bilirubin, Alkaline Phosphatase);
* Coagulopathy;
* Use medications known to affect dopaminergic function, including MAO inhibitors, tetrabenazine, or levodopa;
* Recent (within 3 months) or current treatment with drugs influencing beta cell function or insulin sensitivity (e.g. glucocorticoids, reserpine);
* Have polycystic ovarian syndrome;
* History of movement disorder such as Parkinson's Disease, Huntington's Disease;
* Clinically significant psychiatric disease or history of psychiatric illness such as depression, bipolar disease, anxiety or schizophrenia;
* Current use (within past year) of cocaine, methamphetamine, and/or ecstasy ( MDMA, 34- methylenedioxymethamphetamine;
* Have a recent history of alcohol or substance abuse or dependence;
* Clinically significant cardiovascular disease or clinically significant abnormalities on screening ECG (including but not limited to QTc>450 msec);
* Clinically significant pulmonary, renal or hepatic impairment, or cancer;
* Have clinically significant infectious disease, including AIDS or HIV infection or previous positive test for hepatitis B, hepatitis C, HIV-1, or HIV-2;
* Are women of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using adequate contraception. Women must not be pregnant (negative serum β-HCG at the time of screen) or breastfeeding at screening, and must agree to take appropriate steps not to become pregnant for 30 days following the clinical trial;
* Require medications with a narrow therapeutic window (e.g., warfarin), are receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days;
* Weigh more than the manufacturer-recommended limit for the PET/CT camera being used;
* Any prior participation in other research protocols within the past month that involved radiation, with the exception of plain radiography studies (i.e., chest x-rays); and
* Have received a diagnostic or therapeutic radiopharmaceutical within the past week.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pancreatic uptake and clearance of 18F-AV-133 tracer as determined by SUVR | 0-90 minutes
  SUVR=standard uptake value ratio

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (1):
- Research Site, New York, New York, United States